CLINICAL TRIAL: NCT00757536
Title: Primary Vitrectomy Combined With 360° Endolaser or Encircling Band for Rhegmatogenous Retinal Detachment (V.E.E. Study)
Brief Title: Primary Vitrectomy With Endolaser or Encircling Band for Rhegmatogenous Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Principal Investigator, Dr. Christiane I. Falkner-Radler, principal investigator, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR-3-CI-2008
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Rhegmatogenous Retinal Detachment; Primary Vitrectomy; Encircling Band; Endolaser Treatment
Keywords: Rhegmatogenous retinal detachment; primary vitrectomy; encircling band; endolaser treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Procedure: Encircling Band
- Group 2 (Active Comparator)
  Interventions: Procedure: Endolaser Photocoagulation

INTERVENTIONS:
Procedure: Encircling Band — ppVE and encircling band
  Arms: Group 1
Procedure: Endolaser Photocoagulation — ppVE and endolaser photocoagulation
  Arms: Group 2

SUMMARY:
Comparing primary PPV with 360° endolaser photocoagulation with primary PPV with an encircling band for patients with RRDs.

DETAILED DESCRIPTION:
published

ELIGIBILITY:
Inclusion Criteria:

* Primary rhegmatogenous retinal detachment with or without macula-off detachment phakic or pseudophakic eyes
* Multiple breaks, inferior and posterior located breaks or unclear hole formation
* Proliferative vitreoretinopathy (PVR) stage A and B

Exclusion Criteria:

* Previous retinal detachment surgery
* Giant tears
* PVR stage C
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Retinal redetachment rate | 6 months

SECONDARY OUTCOMES:
Surgery-related complications, patients' comfort, refractive change, visual acuity and optical coherence tomography. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, MD, Study Chair — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery; Christiane I Falkner-Radler, MD, Principal Investigator — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Locations (1):
- The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falkner-Radler CI, Graf A, Binder S. Vitrectomy combined with endolaser or an encircling scleral buckle in primary retinal detachment surgery: a pilot study. Acta Ophthalmol. 2015 Aug;93(5):464-469. doi: 10.1111/aos.12663. Epub 2015 Jan 28. PMID 25626910